CLINICAL TRIAL: NCT02614573
Title: International Normalised Ratio Evaluation by Generalist Practitioners in Full-time Care Establishments for the Elderly: a Pilot Study
Brief Title: International Normalised Ratio Evaluation by Generalist Practitioners in Full-time Care Establishments for the Elderly
Acronym: INR-Cap pilote
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/CS-01; 2015-A01056-43 (Other: ANSM)
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-08

CONDITIONS: Aged; Nursing Homes
Keywords: Dependent; Aged, 80 and over; Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The clinical phases of this study will be held in the nursing home (EHPAD; principal building + 2 annexes) of Pont-Saint-Esprit, located in France. Patients are elderly dependents treated by anti-vitamin K for more than 6 months.
  Interventions: Device: CoagucheckXSR Capillary INR measures

INTERVENTIONS:
Device: CoagucheckXSR Capillary INR measures — We will be using the CoagucheckXSR device for capillary INR measures performed by nurses every 7 days during the 6 months of the study, plus after related intercurrent events.
  If capillary INR is <2 or >3 (with a tolerance of 1.9 to 3.1 given the margin of measurement inaccuracy of the coagulometer), then a classic venous measure is performed. If both tests agree, adaptation of treatment as indicated. If slightly discordant results, then the INR values are considered discordant and the decision to adjust the treatment dose and the next monitoring date for venous INR is made based on the value of the venous INR, according to the predefined protocol. If clinically significant discordance (> 0.3), a venous INR is reperformed within 24 hours and if the discrepancy persists, dose adjustment is made according to the venous INR and the predefined protocol.
  If capillary INR is > 4, then verification by venous measure and refer to general practitioner.
  Other Names: CoagucheckXSR

SUMMARY:
The main objective of this study is to evaluate, for a 6-month observation period, the concordance in terms of clinical decision making concerning therapeutic adjustment as determined by a weekly capillary International Normalised Ratio (INR) monitoring strategy versus the usual strategy in a population of dependent elderly people in nursing homes, treated with anti-vitamin K (AVK).

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

A. Estimate the intra-patient variability of capillary INR measures.

B. Estimate the time spent in the target INR (TTR) window of dependent elderly patients in nursing homes, under AVK treatment, and with a capillary INR monitoring strategy.

C. Estimate the number of venous thromboembolic events and bleeding events over the 6-month observation period.

ELIGIBILITY:
Inclusion Criteria:

* The patient resides at the establishment for the dependent elderly (nursing home (EHPAD)) in Pont-Saint-Esprit, France
* The patient must be insured or beneficiary of a health insurance plan
* The patient treated with vitamin K antagonist for over six months
* The patient must have given his/her informed and signed consent
* For adults under guardianship, the legal guardian must have given free and informed consent and signed the consent

Exclusion Criteria:

* The patient is under judicial protection
* The general practitioner in charge of the patient at the EHPAD does not want to participate in the study
* It is impossible to correctly inform the patient, or his/her legal guardian
* The patient, or his/her legal guardian, refuses to sign the consent
* The patient is participating in another interventional study, or has participated in another interventional study within the past three months
* The patient is in an exclusion period determined by a previous study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08-13 (Actual); Study Completion 2016-08-13 (Actual)

PRIMARY OUTCOMES:
Is the capillary INR concordant with the venous INR ? yes/no | 6 months
  Primary Outcome Measure as stated in protocol: Clinical concordances and clinical discrepancies between the capillary INR and venous INR every time they are concomitant

SECONDARY OUTCOMES:
The number of thromboembolic events per patient | 6 months
The number of bleeding events per patient | 6 months
The number of thromboembolic or bleeding events per patient | 6 months
Coefficient of variation for capillary INR measures per patient | 6 months
Time in therapeutique range (days) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Sikirdji, Interne, Study Director — Centre Hospitalier Universitaire de Nîmes; Jean-François Clape, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- EHPAD de l'Hôpital de Pont Saint Esprit, Pont-Saint-Esprit, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sikirdji C, Costa D, Alonso S, Clape JF, Amouyal M, de Waziere B, Fabbro-Peray P. Assessment of agreement and time in therapeutic range of capillary versus venous international normalised ratio in frail elderly people in a nursing home. Intern Med J. 2019 Nov;49(11):1442-1446. doi: 10.1111/imj.14626. PMID 31713344